CLINICAL TRIAL: NCT03006367
Title: An Open-label, Single Ascending Dose, Pharmacokinetic and Tolerability Study of NFC-1 in Children and Adolescents (Ages 6-17 Years) With Attention Deficit Hyperactivity Disorder
Brief Title: Pharmacokinetic and Tolerability Study of NFC-1 in Subjects Aged 6-17 Years With ADHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDGN-NFC1-ADHD-101
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NFC-1 100 mg (Experimental): Single Dose of NFC-1 100 mg
  Interventions: Drug: NFC-1 100 mg
- NFC-1 200 mg (Experimental): Single Dose of NFC-1 200 mg
  Interventions: Drug: NFC-1 200 mg
- NFC-1 400 mg (Experimental): Single Dose of NFC-1 400 mg
  Interventions: Drug: NFC-1 400 mg
- NFC-1 800 mg (Experimental): Single Dose of NFC-1 800 mg
  Interventions: Drug: NFC-1 800 mg

INTERVENTIONS:
Drug: NFC-1 100 mg
  Other Names: AEVI-001; MDGN-001
  Arms: NFC-1 100 mg
Drug: NFC-1 200 mg
  Other Names: AEVI-001; MDGN-001
  Arms: NFC-1 200 mg
Drug: NFC-1 400 mg
  Other Names: AEVI-001; MDGN-001
  Arms: NFC-1 400 mg
Drug: NFC-1 800 mg
  Other Names: AEVI-001; MDGN-001
  Arms: NFC-1 800 mg

SUMMARY:
This is a open-label, single ascending dose, pharmacokinetic, and tolerability study of NFC-1 in Children and Adolescents (Ages 6-17 Years) with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and parent/legally authorized representative (LAR) are able to speak English fluently and have provided written informed consent, and assent (as applicable) for this study.
2. Subject is 6 to 17 years inclusive at the time of consent/assent.
3. Subject is male, female of non-childbearing potential or non-pregnant, non-lactating female of childbearing potential who agrees to comply with any applicable contraceptive requirements 2 weeks prior to administration of IP and throughout the study.
4. Subject meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD based on a M.I.N.I. International Neuropsychiatric Interview.
5. Subject is considered "healthy". Healthy status is defined by absence of evidence of any active or chronic disease other than their ADHD following a detailed medical and surgical history, a complete physical examination.
6. Subject has the ability to swallow a capsule of investigational product whole.

Exclusion Criteria:

1. Subject has a history of any hematological, hepatic, respiratory, cardiovascular, renal, neurological, or psychiatric disease, gall bladder removal, or current or recurrent disease other than their ADHD.
2. Subject has a current or relevant history of physical or psychiatric illness, or any medical disorder that may require treatment.
3. Subject has a current, controlled or uncontrolled, comorbid psychiatric diagnosis with significant symptoms.
4. Subject is considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation.
5. Subject has used an investigational product, been enrolled in a clinical study including vaccines, or had any changes in eating habits, within 30 days prior to the first dose of investigational product.
6. Subject has a positive screen for alcohol or drugs of abuse, or a positive hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or HIV antibody screen.
7. Subject previously was an adolescent (12-17) who was either a screen failure, or enrolled or participated in this study or another NFC1 clinical study.
8. Subject is currently taking any medication that might confound the results of safety assessments conducted in the study.
9. Subject has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments conducted in the study.
10. Subject is unwilling to discontinue current ADHD medication to participate in the study.
11. Subject has a clinical laboratory abnormality that indicates clinically significant hematologic, hepatobiliary, or renal disease.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2017-02-26 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve (AUC0-24h) | 24 hours of sample collections
Area under the plasma drug concentration-time curve (AUC0-inf) | 28 hours of sample collections
Area under the plasma drug concentration-time curve (AUClast) | 28 hours of sample collections
Terminal Half Life (T½ ) of NFC-1 | 28 hours of sample collections
Maximum Observed Plasma Concentration (Cmax) | 28 hours of sample collections
Time to Maximum Observed Plasma Concentration (Tmax) | 28 hours of sample collections
Apparent first order elimination rate constant (kel) | 28 hours of sample collections
Apparent oral clearance adjusted for bioavailability (CL/F) of NFC-1 | 28 hours of sample collections
Apparent volume of distribution adjusted for bioavailability (Vz/F) of NFC-1 | 28 hours of sample collections

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Meridien Research, Inc., Maitland, Florida
  - QPS-MRA, LLC (Miami Research Associates), Miami, Florida
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glessner JT, Khan ME, Chang X, Liu Y, Otieno FG, Lemma M, Slaby I, Hain H, Mentch F, Li J, Kao C, Sleiman PMA, March ME, Connolly J, Hakonarson H. Rare recurrent copy number variations in metabotropic glutamate receptor interacting genes in children with neurodevelopmental disorders. J Neurodev Disord. 2023 Apr 29;15(1):14. doi: 10.1186/s11689-023-09483-z. PMID 37120522
- [Derived] Slaby I, Hain HS, Abrams D, Mentch FD, Glessner JT, Sleiman PMA, Hakonarson H. An electronic health record (EHR) phenotype algorithm to identify patients with attention deficit hyperactivity disorders (ADHD) and psychiatric comorbidities. J Neurodev Disord. 2022 Jun 11;14(1):37. doi: 10.1186/s11689-022-09447-9. PMID 35690720